CLINICAL TRIAL: NCT03861975
Title: Exploring the Efficacy and Feasibility of the LymphaTech Scanner for Breast Cancer-Related Lymphedema Screening
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Heinz Family Foundation (Unknown)
Responsible Party: Principal Investigator, Alphonse Taghian, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 18-181
Record Dates: First submitted 2019-03-01; First posted 2019-03-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is an interventional, non-therapeutic screening trial comparing two measurement devices cross-sectionally.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast Cancer-Related Lymphedema Measurements (Experimental): Absolute volume of the upper extremities will be assessed using the LymphaTech Scanner and the Perometer.
  Interventions: Other: Breast Cancer-Related Lymphedema Measurements

INTERVENTIONS:
Other: Breast Cancer-Related Lymphedema Measurements — All patients will receive bilateral arm measurements using the LymphaTech Scanner and the Perometer.

SUMMARY:
This research will compare the absolute volumes of the upper extremity using both the LymphaTech Scanner and Perometer in a cohort of patients with a history of invasive or in-situ carcinoma of the breast.

DETAILED DESCRIPTION:
Our trial seeks to assess the efficacy of the LymphaTech Scanner as compared to the Perometer, which is currently used to screen for breast cancer-related lymphedema. The focus of the study is to compare the absolute volumes of the upper-extremity as measured by each device and to compare the time it takes to measure both arms of a patient using each device to assess clinical feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed invasive or in-situ carcinoma of the breast and will undergo unilateral breast cancer surgery
* Age >18 years.
* Ability to understand and the willingness to verbally consent to the trial

Exclusion Criteria:

* History of primary lymphedema.
* Any patient with a current case of cellulitis.
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Participants unable to abduct upper-extremity perpendicular to body or to stand comfortably without aid for several minutes, both of which are necessary to perform a LymphaTech Scan

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-30 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Precision and reliability | 3 years
  To determine whether the LymphaTech scanner is a precise and reliable tool for measuring upper extremity volume changes in patients treated for breast

SECONDARY OUTCOMES:
Measurement Time | 3 years
  To evaluate amount of time it takes to conduct bilateral arm measurements with both the LymphaTech Scanner and Perometer.

CONTACTS AND LOCATIONS:
Overall Officials: Alphonse G. Taghian, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation